CLINICAL TRIAL: NCT04401462
Title: SCORE Trial - Scandinavian Olecranon Research in the Elderly
Brief Title: Scandinavian Olecranon Research in the Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Helsinki University Central Hospital (Other); Oulu University Hospital (Other); Kuopio University Hospital (Other); University Hospital, Linkoeping (Other); Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCORE
Record Dates: First submitted 2020-05-19; First posted 2020-05-26 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Olecranon Fracture
MeSH Terms: conditions — Olecranon Fracture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Operative group (Active Comparator): tension band wiring or plate fixation
  Interventions: Procedure: Tension band wiring or plate fixation
- Non-operative group (Active Comparator): conservative treatment
  Interventions: Behavioral: Sling or a long-arm plaster

INTERVENTIONS:
Procedure: Tension band wiring or plate fixation — Operative fixation of olecranon fracture with either of the methods mentioned in the intervention name
  Arms: Operative group
Behavioral: Sling or a long-arm plaster — Non-operative treatment and progressive range of motion as tolerated. A long-arm plaster will be used, if necessary, for pain relief.
  Arms: Non-operative group

SUMMARY:
This study is designed to study the difference between operative treatment, either with tension band wiring or plate fixation, and conservative treatment of traumatic, displaced olecranon fractures in elderly population in a non-inferiority study setting.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically (standard AP and lateral radiographs) confirmed, displaced (≥2mm dislocation of the joint surface) fracture of the olecranon
* Age of patient is 75 years or over at the time of the injury

Exclusion Criteria:

* A delay more than 2 weeks after traumatic event to the day of intervention
* Mayo type 3 fracture
* Fracture continuation distal to coronoideus
* Other acute fracture or nerve damage of the ipsilateral upper limb
* Old fracture (<6 months) or pseudoarthrosis or unhealed nerve injury of the ipsilateral upper limb
* Open fracture
* Pathological fracture
* History of alcoholism, drug abuse, psychological or other emotional problems likely to jeopardize informed consent
* Patient's inability to understand written and spoken Finnish or Swedish or Danish
* Patient's denial for participation or cognitive incapability to provide consent
* Patient physically unfit for surgery

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
the Disabilities of Arm, Shoulder and Hand (DASH) | 1 year
  Minimum value 0, maximum value 100. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
the Disabilities of Arm, Shoulder and Hand (DASH) | 3 months
  Minimum value 0, maximum value 100. Higher scores mean worse outcome.
Patient Rated Elbow Evaluation (PREE) Finnish, Swedish and Danish versions | 3 and 12 months
  Minimum value 0, maximum value 100. Higher score indicates more pain and functional disability.
Pain, visual analogue scale (VAS) | 3 and 12 months
  Minimum value 0, maximum value 100. Higher scores mean worse outcome ie. more pain.
Satisfaction, visual analogue scale (VAS) | 3 and 12 months
  Minimum value 0, maximum value 100. Higher scores mean worse outcome ie. less satisfactory situation.
Elbow X-rays | post-operatively, 2 weeks, 3 and 12 months
  AP and lateral view.
Range of elbow motion. | 3 and 12 months
  The results are reported in degrees. Measurement is performed to the injured arm.
Comparison of extension strength between injured and healthy elbow. | 12 months
  Both arms are measured elbow flexed 60 and 90 degrees. Power is reported in grams. Measurements are performed in sitting position, back straight.
Adverse events | up to 12 months

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (3):
  - Turku Central University Hospital, Turku, Southwest Finland
  - Hospital Nova, Jyväskylä
  - Tampere University Hospital, Tampere
- Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rantalaiho I, Laaksonen I, Launonen AP, Luokkala T, Flinkkila T, Salmela M, Adolfsson L, Olsen B, Isotalo K, Ryosa A, Aarimaa V; SCORE study group. Scandinavian Olecranon Research in the Elderly (SCORE): protocol for a non-inferiority, randomised, controlled, multicentre trial comparing operative and conservative treatment of olecranon fractures in the elderly. BMJ Open. 2022 Jan 31;12(1):e055097. doi: 10.1136/bmjopen-2021-055097. PMID 35105643